CLINICAL TRIAL: NCT00410280
Title: Allergen Challenge
Brief Title: Study Evaluating the Effects of IMA-638 on Allergen-Induced Airway Responses in Subjects With Mild Atopic Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3174K1-200; B2421001 (Other: Alias Study Number)
Record Dates: First submitted 2006-12-08; First posted 2006-12-12 (Estimated); Results first posted 2014-11-18 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Biological: IMA-638 is a biologic

INTERVENTIONS:
Biological: IMA-638 is a biologic

SUMMARY:
Primary purpose of the protocol is to determine if IMA-638 prevents a mild asthma attack by a subject with mild asthma inhaling an allergen.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* generally healthy, men and women with mild allergic asthma, aged 18 to 60 years
* only asthma med is short-acting bronchodilator used not more than twice weekly
* FEV1 greater than 70% predicted and a demonstrated baseline late response to allergen induction

Exclusion Criteria:

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Canada (3):
  - University of British Columbia, Vancouver, British Columbia
  - McMaster University Medical, Hamilton, Ontario
  - Hopital Laval, Ste-Foy, Quebec

REFERENCES:
- [Derived] Gauvreau GM, Boulet LP, Cockcroft DW, Fitzgerald JM, Carlsten C, Davis BE, Deschesnes F, Duong M, Durn BL, Howie KJ, Hui L, Kasaian MT, Killian KJ, Strinich TX, Watson RM, Y N, Zhou S, Raible D, O'Byrne PM. Effects of interleukin-13 blockade on allergen-induced airway responses in mild atopic asthma. Am J Respir Crit Care Med. 2011 Apr 15;183(8):1007-14. doi: 10.1164/rccm.201008-1210OC. Epub 2010 Nov 5. PMID 21057005
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3174K1-200&StudyName=Study%20Evaluating%20the%20Effects%20of%20IMA-638%20on%20Allergen-Induced%20Airway%20Responses%20in%20Subjects%20with%20Mild%20Atopic%20Asthma

RESULTS

PARTICIPANT FLOW:
Groups:
- IMA-638 2mg/kg: IMA-638 2 milligram/kilogram (mg/kg) subcutaneous injection on Day 1 and 8.
- Placebo: Placebo matched to IMA-638 subcutaneous injection on Day 1 and 8.
Period: Overall Study
Arm/Group | IMA-638 2mg/kg | Placebo
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population (ITT) included all randomized participants who received at least 1 dose administration of the test article.
Groups:
- Total: Total of all reporting groups
Arm/Group | IMA-638 2mg/kg | Placebo | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.14 (6.25) | 32.31 (11.66) | 29.11 (9.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Maximum Percent Drop From Pre-allergen Baseline in Forced Expiratory Volume in 1 Second (FEV1) for Late-Phase Asthma Response (LAR) at Screening
Description: Allergen inhalation test was performed at Screening, Day 14 and 35 to elicit airway responses similar to those that follow natural allergen exposure. FEV1 was the maximal volume of air exhaled in 1 second of a forced expiration from a position of full inspiration. LAR was characterized by a fall in FEV1 of more than or equal to (>=) 15 percent (%) at 3 to 7 hours post-allergen inhalation. Maximum drop in FEV1 relative to the pre-allergen baseline FEV1 between 3 to 7 hours at Screening was reported. Pre-allergen baseline FEV1 was performed in triplicate using spirometry and the best of the 3 values was selected.
Time Frame: Pre-allergen baseline, 3, 4, 5, 6, 7 hours post-allergen inhalation at Screening (Day -14)
Population: ITT population included all randomized participants who received at least 1 dose administration of the test article.
Measure: Mean (Standard Deviation); unit: percent drop
Arm/Group | IMA-638 2mg/kg | Placebo
Number analyzed (Participants) | 14 | 13
percent drop | 27.19 (9.75) | 20.47 (8.12)

2. Primary Outcome: Maximum Percent Drop From Pre-allergen Baseline in Forced Expiratory Volume in 1 Second (FEV1) for Late-Phase Asthma Response (LAR) at Day 14
Description: Allergen inhalation test was performed at Screening, Day 14 and 35 to elicit airway responses similar to those that follow natural allergen exposure. FEV1 was the maximal volume of air exhaled in 1 second of a forced expiration from a position of full inspiration. LAR was characterized by a fall in FEV1 of more than or equal to (>=) 15 percent (%) at 3 to 7 hours post-allergen inhalation. Maximum drop in FEV1 relative to the pre-allergen baseline FEV1 between 3 to 7 hours on Day 14 was reported. Pre-allergen baseline FEV1 was performed in triplicate using spirometry and the best of the 3 values was selected.
Time Frame: Pre-allergen baseline, 3, 4, 5, 6, 7 hours post-allergen inhalation at Day 14
Population: ITT population included all randomized participants who received at least 1 dose administration of the test article.
Measure: Mean (Standard Deviation); unit: percent drop
Arm/Group | IMA-638 2mg/kg | Placebo
Number analyzed (Participants) | 14 | 13
percent drop | 12.84 (10.29) | 19.28 (10.69)
Statistical Analysis 1: Comparison: IMA-638 2mg/kg vs Placebo; Repeated measures analysis of variance (ANOVA) model with fixed effects for treatment, time and interaction between treatment and time, and random effects for participant was used. Point estimate for difference between the treatment groups, corresponding 95 % confidence interval (CI) and p-value were derived from the model; Test type: Superiority or Other; p = 0.0947, ANOVA; Mean Difference (Final Values) = -6.44, 95% CI 2-sided [-14.04 to 1.15]

3. Primary Outcome: Maximum Percent Drop From Pre-allergen Baseline in Forced Expiratory Volume in 1 Second (FEV1) for Late-Phase Asthma Response (LAR) at Day 35
Description: Allergen inhalation test was performed at Screening, Day 14 and 35 to elicit airway responses similar to those that follow natural allergen exposure. FEV1 was the maximal volume of air exhaled in 1 second of a forced expiration from a position of full inspiration. LAR was characterized by a fall in FEV1 of more than or equal to (>=) 15 percent (%) at 3 to 7 hours post-allergen inhalation. Maximum drop in FEV1 relative to the pre-allergen baseline FEV1 between 3 to 7 hours on Day 35 was reported. Pre-allergen baseline FEV1 was performed in triplicate using spirometry and the best of the 3 values was selected.
Time Frame: Pre-allergen baseline, 3, 4, 5, 6, 7 hours post-allergen inhalation at Day 35
Population: ITT population included all randomized participants who received at least 1 dose administration of the test article.
Measure: Mean (Standard Deviation); unit: percent drop
Arm/Group | IMA-638 2mg/kg | Placebo
Number analyzed (Participants) | 14 | 13
percent drop | 11.32 (9.39) | 15.56 (10.45)
Statistical Analysis 1: Comparison: IMA-638 2mg/kg vs Placebo; Repeated measures ANOVA model with fixed effects for treatment, time and interaction between treatment and time, and random effects for participant was used. Point estimate for difference between the treatment groups, corresponding 95% CI and p-value were derived from the model; Test type: Superiority or Other; p = 0.2673, ANOVA; Mean Difference (Final Values) = -4.24, 95% CI 2-sided [-11.84 to 3.35]

4. Secondary Outcome: Area Under the Percent Drop in Forced Expiratory Volume in 1 Second Curve (AUC FEV1) From Time 3 to 7 Hours for Late-Phase Asthma Response (LAR)
Description: Allergen inhalation test was performed at Screening, Day 14 and 35 to elicit airway responses similar to those that follow natural allergen exposure. FEV1 was the maximal volume of air exhaled in 1 second of a forced expiration from a position of full inspiration. LAR was characterized by a fall in FEV1 of >=15% at 3 to 7 hours post-allergen inhalation. Area under the percent drop in FEV1 relative to the pre-allergen baseline FEV1 from 3 to 7 hours was computed using the linear trapezoidal rule. Pre-allergen baseline FEV1 was performed in triplicate using spirometry and the best of the 3 values was selected.
Time Frame: Pre-allergen baseline, 3, 4, 5, 6, 7 hours post-allergen inhalation at Screening (Day -14), Day 14, 35
Population: ITT population included all randomized participants who received at least 1 dose administration of the test article.
Measure: Mean (Standard Deviation); unit: Percent drop*hour
Arm/Group | IMA-638 2mg/kg | Placebo
Number analyzed (Participants) | 14 | 13
Percent drop*hour
  Screening | 57.57 (24.26) | 55.64 (27.78)
  Day 14 | 25.48 (29.49) | 49.28 (32.66)
  Day 35 | 21.94 (21.27) | 39.11 (37.46)
Statistical Analysis 1: Comparison: IMA-638 2mg/kg vs Placebo; Day 14: Repeated measures ANOVA model with fixed effects for treatment, time and interaction between treatment and time, and random effects for participant was used. Point estimate for difference between the treatment groups, corresponding 95% CI and p-value were derived from the model; Test type: Superiority or Other; p = 0.0391, ANOVA; Mean Difference (Final Values) = -23.80, 95% CI 2-sided [-46.35 to -1.24]
Statistical Analysis 2: Comparison: IMA-638 2mg/kg vs Placebo; Day 35: Repeated measures ANOVA model with fixed effects for treatment, time and interaction between treatment and time, and random effects for participant was used. Point estimate for difference between the treatment groups, corresponding 95% CI and p-value were derived from the model; Test type: Superiority or Other; p = 0.1326, ANOVA; Mean Difference (Final Values) = -17.17, 95% CI 2-sided [-39.72 to 5.39]

5. Secondary Outcome: Maximum Percent Drop From Pre-allergen Baseline in Forced Expiratory Volume in 1 Second (FEV1) for Early-Phase Asthma Response (EAR) at Screening, Day 14 and 35
Description: Allergen inhalation test was performed at Screening, Day 14 and 35 to elicit airway responses similar to those that follow natural allergen exposure. FEV1 was the maximal volume of air exhaled in 1 second of a forced expiration from a position of full inspiration. EAR was characterized by a fall in FEV1 >=20% at 0 to 3 hours post-allergen inhalation. Maximum drop in FEV1 relative to the pre-allergen baseline FEV1 between 0 to 3 hours was reported. Pre-allergen baseline FEV1 was performed in triplicate using spirometry and the best of the 3 values was selected.
Time Frame: Pre-allergen baseline, 10, 20, 30, 45, 60, 90, 120, 180 minutes post-allergen inhalation Screening, Day 14, 35
Population: ITT population included all randomized participants who received at least 1 dose administration of the test article.
Measure: Mean (Standard Deviation); unit: percent drop
Arm/Group | IMA-638 2mg/kg | Placebo
Number analyzed (Participants) | 14 | 13
percent drop
  Screening | 33.23 (6.26) | 34.40 (8.51)
  Day 14 | 20.40 (14.98) | 30.15 (13.57)
  Day 35 | 22.76 (13.51) | 26.82 (13.56)
Statistical Analysis 1: Comparison: IMA-638 2mg/kg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0423, ANOVA; Mean Difference (Final Values) = -9.76, 95% CI 2-sided [-19.16 to -0.35]
Statistical Analysis 2: Comparison: IMA-638 2mg/kg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.3902, ANOVA; Mean Difference (Final Values) = -4.06, 95% CI 2-sided [-13.46 to 5.35]

6. Secondary Outcome: Area Under the Percent Drop in Forced Expiratory Volume in 1 Second Curve (AUC FEV1) From Time 0 to 3 Hours for Early-Phase Asthma Response (EAR)
Description: Allergen inhalation test was performed at Screening, Day 14 and 35 to elicit airway responses similar to those that follow natural allergen exposure. FEV1 was the maximal volume of air exhaled in 1 second of a forced expiration from a position of full inspiration. EAR was characterized by a fall in FEV1 >=20% at 0 to 3 hours post-allergen inhalation. Area under the percent drop in FEV1 relative to the pre-allergen baseline FEV1 from 0 to 3 hours at each visit was computed using the linear trapezoidal rule. Pre-allergen baseline FEV1 was performed in triplicate using spirometry and the best of the 3 values was selected.
Time Frame: Pre-allergen baseline, 10, 20, 30, 45, 60, 90, 120, 180 minutes post-allergen inhalation Screening, Day 14, 35
Population: ITT population included all randomized participants who received at least 1 dose administration of the test article.
Measure: Mean (Standard Deviation); unit: percent drop*hour
Arm/Group | IMA-638 2mg/kg | Placebo
Number analyzed (Participants) | 14 | 13
percent drop*hour
  Screening | 45.37 (15.03) | 50.39 (24.09)
  Day 14 | 21.51 (23.20) | 40.56 (26.62)
  Day 35 | 25.75 (18.21) | 38.94 (24.42)
Statistical Analysis 1: Comparison: IMA-638 2mg/kg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0302, ANOVA; Mean Difference (Final Values) = -19.05, 95% CI 2-sided [-36.21 to -1.90]
Statistical Analysis 2: Comparison: IMA-638 2mg/kg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.1289, ANOVA; Mean Difference (Final Values) = -13.19, 95% CI 2-sided [-30.34 to 3.97]

7. Secondary Outcome: Change From Pre-allergen Challenge in Provocative Concentration of Methacholine Causing a 20% Fall in FEV1 (PC20) to Post-allergen Challenge For Screening, Day 14 and 35 Challenge
Description: Methacholine inhalation test was performed to determine airway hyper-reactivity using provocative concentration 20 (PC20). PC20 was the lowest concentration of methacholine at which participant had 20% decrease from baseline in FEV1. Pre-allergen challenge methacholine inhalation test was performed 1 day prior to the allergen challenge and post-allergen challenge methacholine inhalation test was performed 1 day after to the allergen challenge (that is, pre- and post-allergen methacholine inhalation test was conducted on Day -15 and -13 for Screening allergen challenge, Day 13 and 15 for Day 14 allergen challenge and Day 34 and 36 for Day 35 allergen challenge, respectively). For each methacholine inhalation test, baseline FEV1 was defined as the lowest value among the triplicate readings taken after administration of the diluent (saline administration). Difference between post-allergen challenge and pre-allergen challenge was expressed as log2 (post-allergen PC20 - pre-allergen PC20).
Time Frame: Day -15, -13 for Screening (Day -14) challenge; Day 13, 15 for Day 14 challenge; Day 34, 36 for Day 35 challenge
Population: ITT population included all randomized participants who received at least 1 dose administration of the test article.
Measure: Mean (Standard Deviation); unit: Log2 milligram/milliliter (log2 mg/mL)
Arm/Group | IMA-638 2mg/kg | Placebo
Number analyzed (Participants) | 14 | 13
Log2 milligram/milliliter (log2 mg/mL)
  Screening | -1.37 (0.74) | -1.47 (1.72)
  Day 14 | -0.63 (1.20) | -0.63 (1.28)
  Day 35 | -0.71 (0.97) | -0.43 (0.72)
Statistical Analysis 1: Comparison: IMA-638 2mg/kg vs Placebo; Screening: Mixed model with fixed effects for treatment, time and interaction between treatment and time, and random effects for participants was used. Point estimate for difference between the treatment groups, corresponding 95% CI and p-values were derived from the model; Test type: Superiority or Other; p = 0.8469, Mixed Models Analysis; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.79 to 0.96]
Statistical Analysis 2: Comparison: IMA-638 2mg/kg vs Placebo; Day 14: Mixed model with fixed effects for treatment, time and interaction between treatment and time, and random effects for participants was used. Point estimate for difference between the treatment groups, corresponding 95% CI and p-values were derived from the model; Test type: Superiority or Other; p = 0.9995, Mixed Models Analysis; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.86 to 0.86]
Statistical Analysis 3: Comparison: IMA-638 2mg/kg vs Placebo; Day 35: Mixed model with fixed effects for treatment, time and interaction between treatment and time, and random effects for participants was used. Point estimate for difference between the treatment groups, corresponding 95% CI and p-values were derived from the model; Test type: Superiority or Other; p = 0.5280, Mixed Models Analysis; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-1.14 to 0.59]

8. Secondary Outcome: Change From Baseline in Total and Differential Sputum Cell Counts at Day 14 and 35
Description: The collected sputum was planned to be analyzed for epithelial cells, eosinophils, lymphocytes, neutrophils, metachromatic cells, or macrophages counts. Sputum induction was to be performed after each methacholine challenge and at 7 hours after each allergen inhalation challenge.
Time Frame: Baseline, Day 14, 35
Population: Data was not analyzed because the study was stopped early after interim analysis and only safety and key efficacy analyses were performed.
Arm/Group | IMA-638 2mg/kg | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Allergen Specific and Total Immunoglobulin E (IgE) Count at Baseline
Description: The baseline for the outcome measure was defined as the last post-dose measurement obtained prior to the allergen challenge within a given challenge triad (planned on day 13 and 34). The challenge triad included pre-allergen methacholine inhalation challenge, allergen inhalation challenge, and post-allergen methacholine inhalation challenge. Results are reported for total IgE count.
Time Frame: Baseline
Population: ITT population included all randomized participants who received at least 1 dose administration of the test article. Allergen-specific IgE was not analyzed because the study was stopped early after interim analysis and only safety and key efficacy analyses were performed.
Measure: Mean (Standard Deviation); unit: kilo unit/liter (kU/L)
Arm/Group | IMA-638 2mg/kg | Placebo
Number analyzed (Participants) | 14 | 13
kilo unit/liter (kU/L) | 259.7 (395.8) | 179.8 (204.7)

10. Secondary Outcome: Change From Baseline in Allergen Specific and Total Immunoglobulin E (IgE) Count at Day 13, 34, 56, 112 and 168
Description: The baseline for the outcome measure was defined as the last post-dose measurement obtained prior to the allergen challenge (planned on Day 13 and 34). Results are reported for total IgE count.
Time Frame: Baseline, Day 13, 34, 56, 112, 168
Population: ITT population. Here, "n" signifies participants evaluated for this measure at the specified time point for each arm. Allergen-specific IgE was not analyzed because the study was stopped early after interim analysis and only safety and key efficacy analyses were performed.
Measure: Mean (Standard Error); unit: kU/L
Arm/Group | IMA-638 2mg/kg | Placebo
Number analyzed (Participants) | 14 | 13
kU/L
  Change at Day 13 (n=14, 13) | 29.1 (23.1) | -4.4 (10.9)
  Change at Day 34 (n=14, 13) | 37.4 (43.9) | 1.5 (8.4)
  Change at Day 56 (n=13, 13) | 4.2 (8.6) | -14.2 (13.8)
  Change at Day 112 (n=13, 13) | -9.2 (21.9) | -32.0 (16.3)
  Change at Day 168 (n=14, 13) | -40.0 (55.6) | -12.2 (31.6)

11. Secondary Outcome: Total Blood Eosinophil Counts at Baseline
Description: The baseline for the outcome measure was defined as the last post-dose measurement obtained prior to the allergen challenge (planned on day 13 and 34).
Time Frame: Baseline
Population: ITT population included all randomized participants who received at least 1 dose administration of the test article.
Measure: Mean (Standard Deviation); unit: 10^9 cells/Liter
Arm/Group | IMA-638 2mg/kg | Placebo
Number analyzed (Participants) | 14 | 13
10^9 cells/Liter | 0.276 (0.140) | 0.315 (0.469)

12. Secondary Outcome: Change From Baseline in Total Blood Eosinophil Counts at Day 8, 13, 21, 34, 56, 84 and 168
Description: as for outcome 11
Time Frame: Baseline, Day 8, 13, 21, 34, 56, 84, 168
Population: ITT population included all randomized participants who received at least 1 dose administration of the test article. Here, "n" signifies participants evaluated for this measure at the specified time point for each arm.
Measure: Mean (Standard Error); unit: 10^9 cells/Liter
Arm/Group | IMA-638 2mg/kg | Placebo
Number analyzed (Participants) | 14 | 13
10^9 cells/Liter
  Change at Day 8 (n=14,13) | 0.051 (0.039) | -0.112 (0.090)
  Change at Day 13 (n=14, 13) | 0.089 (0.044) | -0.056 (0.091)
  Change at Day 21(n=14, 13) | 0.060 (0.062) | -0.008 (0.035)
  Change at Day 34 (n=14, 13) | 0.026 (0.042) | -0.022 (0.039)
  Change at Day 56 (n=12, 13) | 0.023 (0.051) | -0.128 (0.072)
  Change at Day 84 (n=0, 1) | NA (NA) — Data was not presented because none of the participants were evaluable at Day 84 for this reporting arm. | 0.030 (NA) — Standard Error could not been estimated as single participant was evaluable for this reporting arm.
  Change at Day 168 (n=14, 13) | -0.007 (0.051) | -0.141 (0.138)

13. Secondary Outcome: Blood Levels of Interleukin-13 (IL-13)
Time Frame: Screening, baseline, Day 1, 8, 14, 21, 35, 56, 84, 112, 140, 168
Population: Data for this outcome measure was not analyzed because the study was stopped early after interim analysis and only safety and key efficacy analyses were performed.
Arm/Group | IMA-638 2mg/kg | Placebo
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Messenger Ribonucleic Acid (mRNA) Gene Expression in Sputum and Blood
Description: Sputum induction was performed after each methacholine challenge and at hour 7 after each allergen inhalation challenge. The baseline for this outcome measure was defined as the last value prior to dosing.
Time Frame: Screening (Day-13, -14, -15), Day 1, 13, 14, 15, 34, 35, 36, 112
Population: as for outcome 13
Arm/Group | IMA-638 2mg/kg | Placebo
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Protein Expression in Sputum and Blood
Description: as for outcome 14
Time Frame: Screening (Day-13, -14, -15), Day 1, 13, 14, 15, 34, 35, 36, 112
Population: Data for this outcome measure w as not analyzed because the study w as stopped early after interim analysis and only safety and key efficacy analyses w ere performed.
Arm/Group | IMA-638 2mg/kg | Placebo
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) for IMA-638
Time Frame: Day 1, 8, 14, 21, 35, 56, 84, 112, 140, 168
Population: Evaluable population included all randomized participants who received at least 1 dose administration of the test article and had evaluable pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: microgram/milliliter(mcg/mL)
Arm/Group | IMA-638 2mg/kg
Number analyzed (Participants) | 14
microgram/milliliter(mcg/mL) | 30.5 (6.4)

17. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) for IMA-638
Time Frame: Day 1, 8, 14, 21, 35, 56, 84, 112, 140, 168
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IMA-638 2mg/kg
Number analyzed (Participants) | 14
days | 8.5 (4.4)

18. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] for IMA-638
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUC0-t).
Time Frame: Day 1, 8, 14, 21, 35, 56, 84, 112, 140, 168
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: microgram*hour/milliliter (mcg*hr/mL)
Arm/Group | IMA-638 2mg/kg
Number analyzed (Participants) | 14
microgram*hour/milliliter (mcg*hr/mL) | 32259.13 (6255.88)

19. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] for IMA-638
Description: AUC (0 - ∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: Day 1, 8, 14, 21, 35, 56, 84, 112, 140, 168
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: mcg*hr/mL
Arm/Group | IMA-638 2mg/kg
Number analyzed (Participants) | 14
mcg*hr/mL | 32609.32 (6369.46)

20. Secondary Outcome: Serum Decay Half-Life (t1/2) for IMA-638
Description: Serum decay half-life is the time measured for the serum concentration to decrease by one half.
Time Frame: Day 1, 8, 14, 21, 35, 56, 84, 112, 140, 168
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IMA-638 2mg/kg
Number analyzed (Participants) | 14
days | 25.1 (4.7)

21. Secondary Outcome: Number of Participants With Antibodies to IMA-638
Time Frame: Baseline up to Day 168
Population: ITT population included all randomized participants who received at least 1 dose administration of the test article.
Measure: Number; unit: participants
Arm/Group | IMA-638 2mg/kg | Placebo
Number analyzed (Participants) | 14 | 13
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | IMA-638 2mg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 7/14 | 8/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IMA-638 2mg/kg (N=14) | Placebo (N=13)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Injection site bruising (General disorders) | 0 | 1
Injection site erythema (General disorders) | 1 | 0
Injection site paresthesia (General disorders) | 0 | 1
Injection site swelling (General disorders) | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 2 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1
Neck injury (Injury, poisoning and procedural complications) | 0 | 1
Procedural dizziness (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Syncope vasovagal (Nervous system disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was stopped early due to futility of the interim efficacy analysis results. Hence, only safety results and key efficacy results were presented for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.